CLINICAL TRIAL: NCT00426322
Title: Efficacy of Sinus Floor Augmentation Using Large (1-2mm) or Small (0.25-1mm) Bovine Bone Mineral Particles (Bio-Oss®): A Comparative Histomorphometric Clinical Study
Brief Title: Efficacy of Sinus Floor Augmentation Using Large or Small Bovine Bone Mineral.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Lior Shapira, Head of periodontal department, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: shapiral-HMO-CTIL
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Sinus Graft
Keywords: maxillary sinus augmentation; bone graft; bovine bone mineral; dental implants

ARMS (2):
- 1 (Active Comparator): small particles
  Interventions: Device: bovine bone mineral particles (Bio-Oss®)
- 2 (Active Comparator): large particles
  Interventions: Device: bovine bone mineral particles (Bio-Oss®)

INTERVENTIONS:
Device: bovine bone mineral particles (Bio-Oss®) — bovine bone mineral particles used for sinus augmentation prior to dental implant placement
  Other Names: bovine bone mineral particles (Bio-Oss®) small particles; bovine bone mineral particles (Bio-Oss®) large particles

SUMMARY:
The aim of this clinical study is to compare the amount of newly formed bone after bone augmentation with Bio-Oss® (BO) 0.25-1 mm vs. Bio-Oss® (BO) 1-2 mm in the sinus floor augmentation procedure bilaterally in 8 patients.

Hypothesis:

There is no difference in the relative amount of newly formed bone plus BO between the large (1-2 mm) and small (0.25 - 1 mm) granules.

DETAILED DESCRIPTION:
the use of bovine bone mineral particles (Bio-Oss®)in sinus floor augmentation is well established. bovine bone mineral is an oseoconductive material which serves as a space maintainer and a scaffold for bone augmentation. the commercial product is manufactured in two different particles sizes, "large"1-2 mm, and "small"0.25-1 mm.

Comparison: the histologic characteristics of augmented bone after the use of Bio-Oss® (BO) with particle size of 0.25-1 mm vs. Bio-Oss® (BO)with particle size of 1-2 mm.

ELIGIBILITY:
Inclusion Criteria:

* The patients included in this study are over 18 year old men and women.
* The patient must be a candidate for sinus floor augmentation.
* The patient is able to comply with the study-related procedures such as exercising good oral hygiene and attending all follow-up procedures.
* The patient is able to fully understand the nature of the proposed surgery and is able to provide a signed informed consent.

Exclusion Criteria:

* Pregnant women.
* People who smoke more than 10 cigarettes a day.
* Alcohol and drug abusers.
* People suffering from uncontrolled diabetes, severe osteoporosis, rheumatic arthritis, precancer or neoplastic lesions of oral cavity.
* The patient is nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
the relative amount of mineralised tissue (=newly formed bone plus BO) | 20 monthes

SECONDARY OUTCOMES:
Relative amount of newly formed bone, graft residues, bone marrow, residual bone and connective tissue. | 20 monthes
Clinical parameters: | 32 monthes
complications during surgery related to the material. | 20 monthes
post-operative complications. | 20 monthes
Max torque for implant insertion. | 20 monthes
short-term implant survival (up to one year post loading) | 32 monthes

CONTACTS AND LOCATIONS:
Overall Officials: Lior Shapira, PhD, DMD, Principal Investigator — department of periodontology, Hadassah Medical Organization; Tali Chackartchi, DMD, Study Director — department of periodontology,Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel